CLINICAL TRIAL: NCT06716567
Title: Maternal Determinants of Immunity to Influenza (MADI-01)
Brief Title: Maternal Determinants of Immunity to Influenza
Acronym: MADI-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Nicolas Dauby, Clinical Professor, Infectious Disease Department, Centre Hospitalier Universitaire Saint Pierre
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B762020201013
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Vaccination; Infection; Maternal-Fetal Relations; Influenza; Immunoglobulins
MeSH Terms: conditions — Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Pregnant women and non-pregnant women are recruited in parallel.
Who Masked: Outcomes Assessor
Masking Description: Researchers analyzing the immunological outcomes are blinded to the groups of the subjects (pregnant vs non-pregnant).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women (Active Comparator): Pregnant women receive one dose of influenza-containing vaccine during pregnancy.
  Interventions: Biological: Influenza vaccine
- Non-pregnant women (Active Comparator): Non-pregnant women receive one dose of influenza-containing vaccine.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Alpharix-Tetra®, Vaxigrip Tetra® and Influvac Tetra® were used as influenza vaccines in the 2020-2021, 2021-2022, and 2022-2023 seasons respectively.

SUMMARY:
The overall objective of the project is to determine the impact of pregnancy on the response to influenza immunization.

DETAILED DESCRIPTION:
The study compares immune responses to influenza vaccination between a group of pregnant women and a group of non-pregnant controls women. Specifically, the study has three aims:

1. To compare the quality of antibodies induced by influenza immunization in pregnant and non-pregnant women;
2. To identify immune predictors of vaccine responses in pregnant women and compare them to the determinants of vaccine responses in non-pregnant women;
3. To identify immune predictors of the transfer of maternal antibodies to the newborn following influenza immunization during pregnancy;

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and under 40 years.

Exclusion Criteria:

* Grade III/IV anemia
* Human Immunodeficiency Virus (HIV) infection
* Active bacterial infection
* Opportunistic infection (Tuberculosis, cytomegalovirus (CMV), toxoplasmosis, etc)
* Inability to understand the nature and extent of the study and the procedures required
* Current or recent use of immunosuppressive drugs (corticosteroids, anti-tumor necrosis factors (anti-TNF), methotrexate, etc)
* Active neoplasia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Haemagglutination Inhibition Assay titre | 28 days post vaccination
  Haemagglutination Inhibition Assay (HAI) titres are used to measure responses to relevant influenza strains. The HAI method exploits the property of the influenza virus to haemagglutinate red blood cells. HAI titres are determined as the highest serum dilution inhibiting haemagglutination. An HAI titre of >=40 is considered protective in adults.
  HAI titres will be measured in :
  * Pregnant women
  * Non-pregnant women
Haemagglutination Inhibition Assay titre | At delivery
  Haemagglutination Inhibition Assay (HAI) titres are used to measure responses to relevant influenza strains. The HAI method exploits the property of the influenza virus to haemagglutinate red blood cells. HAI titres are determined as the highest serum dilution inhibiting haemagglutination. An HAI titre of >=40 is considered protective in adults.
  HAI titres will be measured in :
  * Pregnant women
  * In umbilical cord blood

SECONDARY OUTCOMES:
Haemagglutination inhibition assay titre | up to 11 months after vaccination
  Haemagglutination Inhibition Assay (HAI) titres are used to measure responses to relevant influenza strains. The HAI method exploits the property of the influenza virus to haemagglutinate red blood cells. HAI titres are determined as the highest serum dilution inhibiting haemagglutination. An HAI titre of >=40 is considered protective in adults.
  HAI titres will be measured in :
  * Pregnant women: at day of vaccination, day 7 post-vaccination, day 28 post-vaccination, at delivery, week 6 and 12 post-delivery
  * Non-pregnant women: at day of vaccination, day 7, day 28, and Month 6 post-vaccination
Micro neutralization assay titre | up to 11 months after vaccination
  Micro neutralization assay (MNA) titres are measured on serum samples with detectable HAI titres to determine cross reactivity to related virus strains. This method assesses the ability of serum antibodies to prevent virus from infecting a single layer of cells in a micro titre plate.
  MNA titres will be measured in :
  * Pregnant women: at day of vaccination, day 7 post-vaccination, day 28 post-vaccination, at delivery, week 6 and 12 post-delivery
  * Non-pregnant women: at day of vaccination, day 7, day 28, and Month 6 post-vaccination
Influenza virus specific IgG titre | up to 11 month after vaccination
  IgG titres specific to influenza virus Hemagglutinin (HA) and Neuraminidase (NA) are measured using conventional Enzyme-linked immunosorbent assay (ELISA) methods. The Enzyme-Linked Lectin Assay (ELLA) is used for detection of NA-specific antibodies only, using reverse genetics viruses with irrelevant HA to ensure only NA antibodies are measured. ELLA is an ELISA variant but adapted to measure the concentration of antibody to NA, determining the amount of sialic acid cleaved from fetuin.
  IgG titres specific to Influenza Antigens will be assessed by ELISA and ELLA in:
  * Pregnant women: at day of vaccination, day 7 post-vaccination, day 28 post-vaccination, at delivery, week 6 and 12 post-delivery
  * Non-pregnant women: at day of vaccination, day 7, day 28, and Month 6 post-vaccination
Influenza virus specific IgG antibody avidity | up to 11 months after vaccination
  IgG avidity will be measured using chaotropic salts.
  IgG avidity will be assessed in :
  * Pregnant women: at day of vaccination, day 7 post-vaccination, day 28 post-vaccination, at delivery, week 6 and 12 post-delivery
  * Non-pregnant women: at day of vaccination, day 7, day 28, and Month 6 post-vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF